CLINICAL TRIAL: NCT05018260
Title: Attention Bias Modification Versus Attention Control in Treatment of Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAUAttentionControl
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Social Anxiety Disorder (Social Phobia); Social Anxiety; Social Anxiety Disorder
Keywords: social anxiety; social phobia; attention bias modification; attention control
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: particiapants, investigators and outcome assessors are blind to allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GCMRT (Experimental): Attention bias modification: participants will receive gaze-contingent feedback according to their viewing patterns on disgusted and neutral faces
  Interventions: Behavioral: Attention Bias Modification
- attention control (Experimental): Attention control modification: participants will receive gaze-contingent feedback according to their viewing patterns on rounded and sharp geometric shapes
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Attention Bias Modification — Feedback according to participants' viewing patterns, in order to modify their attention bias to threat
  Arms: GCMRT
Behavioral: Attention Control — Feedback according to participants' viewing patterns, in order to strengthen their attention control
  Arms: attention control

SUMMARY:
The purpose of this study is to compare the clinical efficacy of treatment using gaze contingent music reward therapy (GC-MRT) with attention control treatment based on a similar paradigm, for social anxiety disorder (SAD)

DETAILED DESCRIPTION:
This study examines the possibility that the effectiveness shown for GC-MRT in the treatment of SAD leans on attention control rather than bias modification. Therefore half of the participants will receive the classic GC-MRT course of treatment while the other half a version of the task with non-emotional stimuli (geometric shapes).

ELIGIBILITY:
Inclusion Criteria:

* A signed consent form
* Men and women between the ages of 18 and 65.
* Meeting a current diagnosis of Social Anxiety Disorder (SP) according to the DSM-IV.
* SP as the primary diagnosis: In cases of co-morbidity, SP will be deemed as the most distressing and clinically significant condition among the co-morbid disorders.
* No current pharmaco-therapy.

Exclusion Criteria:

* A diagnosis of psychotic or bipolar disorders.
* A diagnosis of a neurological disorder (i.e., epilepsy, brain injury).
* Drug or alcohol abuse.
* Any current pharmacological treatment.
* Any current psychotherapeutic treatment.
* Change in treatment during the study.
* Poor judgment capacity (i.e., children under 18 and special populations).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline - the Liebowitz Social Anxiety Scale (LSAS) - Diagnostic Interview scores | at baseline, one week after end of intervention
  The Liebowitz Social Anxiety Scale (LSAS) is a 24-item scale, each item corresponding to a situation selected on the basis of clinical experience. Each item is rated on a severity scale ranging from 0 to 3 with regard to the passing week, measuring separately two components of social anxiety, specifically, fear/anxiety and avoidance of social interaction and performance situations. The minimum and maximum values of the LSAS total score are 0 and 144, respectively, with higher scores mean worse outcome. Although the assessor may request and ask for further detail and adjust the rating based on clinical experience, this option is not often exercised, and inter-rater agreement is not considered to be a relevant concern.

SECONDARY OUTCOMES:
Change from baseline - the Social Phobia Inventory scores | at baseline, one week after end of intervention
  This is a 17-item self-report measure of social anxiety evaluating fear, avoidance and physiological discomfort. Each item is rated on scale ranging from 0 to 4 with a total score ranging from 0 to 68. Higher scores mean worse outcome.
Clinical Global Impression | at baseline, one week after end of intervention
  A global measure of clinician impression improvement and severity of illness, ranging from 1 to 7. Higher scores mean worse outcome.

OTHER OUTCOMES:
Change from baseline -Attention Control Scale- ACS | at baseline, one week after end of intervention
  The Attention Control Scale (ACS) assesses attention control, using 20 items rated from 1 to 4. The total score ranging from 20 to 80, with higher scores mean better outcome.
Change from baseline - Patient Health Questionnaire- PHQ9 | at baseline, one week after end of intervention
  The Patient Health Questionnaire (PHQ9) assesses depressive symptoms using a self-report, 9 question questionnaire. Items are rated on a scale of 0-3 representing the frequency of depressive symptoms over the past 2 weeks. Scores range between 0 to 27, with higher scores mean worse outcome.
Viewing patterns on disgusted and neutral faces, and round/sharp shapes< representing attention bias. | at baseline, one week after end of intervention
  gaze patterns measured using an established eye tracking task, measuring dwell time on different types of stimuli within a 4X4 matrix.
reaction times on the Flanker task, representing attention control | at baseline, one week after end of intervention
  attention control will be measured using the established Flanker test, to assess change from baseline following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No